CLINICAL TRIAL: NCT04694586
Title: A Prospective Multicenter Phase II-study: Pharmacokinetics and Safety of High-Dose Rifampicin and Pyrazinamide in a Shorter Tuberculosis Treatment Compared With Standardized Treatment in Patients With Mild to Moderate Pulmonary TB
Brief Title: Drug Exposure and Safety of a Shorter Tuberculosis Treatment Based on High-Dose Rifampicin and Pyrazinamide
Acronym: HIGHSHORT-RP
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Suspended 15th of Nov 2023 due to conditions affecting recruitment process.
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Katarina Niward, Principal Investigator, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-003721-25
Record Dates: First submitted 2020-11-23; First posted 2021-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Tuberculosis, Pulmonary
Keywords: Drug-susceptible pulmonary tuberculosis; Rifampicin; Pyrazinamide; Shorter tuberculosis treatment; Pharmacokinetics/Pharmacodynamics; PK/PD; TB; Adverse event
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Rifampin; Pyrazinamide; Isoniazid; Protons; Ethambutol

STUDY DESIGN:
Intervention Model Description: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-dose rifampicin and pyrazinamide (Experimental): rifampicin 35 mg/kg for 4 months provided as a combination of fixed drug combination tablets (HRZE for 8 weeks and HR Week 9-16) and single drug tablets of rifampicin (R)
  AND
  pyrazinamide 40 mg/kg the first 2 months provided as a combination of fixed drug combination tablets (HRZE) and single drug tablets of pyrazinamide (Z)
  fixed drug combination tablets are: isoniazid 75 mg + rifampicin 150 mg + pyrazinamide 400 mg + ethambutol 275 mg (HRZE) combination tablets for 8 weeks AND isoniazid 75 mg + rifampicin 150 mg (HR) combination tablets for Weeks 9 to 16 (total treatment duration 4 months)
  Interventions: Drug: rifampicin; Drug: pyrazinamide; Drug: HRZE; Drug: HR
- Standardized TB treatment (No Intervention): isoniazid 75 mg + rifampicin 150 mg + pyrazinamide 400 mg + ethambutol 275 mg (HRZE) combination tablets for 8 weeks AND isoniazid 75 mg + rifampicin 150 mg (HR) combination tablets for Weeks 9-26 (total treatment duration 6 months)

INTERVENTIONS:
Drug: rifampicin — rifampicin 35 mg/kg
  Other Names: rifampin; rimactan; R
  Arms: High-dose rifampicin and pyrazinamide
Drug: pyrazinamide — pyrazinamide 40 mg/kg
  Other Names: Z
  Arms: High-dose rifampicin and pyrazinamide
Drug: HRZE — isoniazid 75 mg + rifampicin 150 mg + pyrazinamide 400 mg + ethambutol 275 mg combination tablets
  Other Names: isoniazid; H; rifampicin; R; pyrazinamide; Z; ethambutol; E
  Arms: High-dose rifampicin and pyrazinamide
Drug: HR — isoniazid 75 mg + rifampicin 150 mg combination tablets
  Other Names: isoniazid; H; rifampicin; R
  Arms: High-dose rifampicin and pyrazinamide

SUMMARY:
Tuberculosis (TB) treatment is long and complex with the risk of poor treatment adherence and treatment failure. Several attempts to shorten treatment of drug-susceptible TB have been unsuccessful. However, recent data support a shortened regimen for mild and moderate pulmonary TB and simultaneous optimization of rifampicin (RIF) and pyrazinamide (PZA).

This phase II clinical study aim to investigate a strategy to shorten TB treatment by exploring safety and drug exposure of a high-dose sterilizing TB regimen.

DETAILED DESCRIPTION:
In five sites in Sweden (Linköping, Norrköping, Jönköping, Kalmar and Stockholm), 40 consenting adult patients with mild to moderate drug-susceptible pulmonary TB will be recruited. The term Actual Study Start Date (stated 23rd of November 2020) refers to when the study opened for recruitment and this date will be updated once the first patient is enrolled in the trial.

The study participants are randomized to receive either 6-month standardized TB treatment (n=10) or a 4-month regimen (n=30) of rifampicin (RIF) 35 mg/kg and isoniazid (INH) 5 mg/kg complemented the first 8 weeks by pyrazinamide (PZA) 40 mg/kg and ethambutol (EMB) 15-20 mg/kg.

First-line drug concentration is determined at 0, 1, 2, 4, 6, 8, 12 and 24 h Day 1 and Week 2 and potential side effects thoroughly monitored throughout the study.

Early bactericidal activity (EBA) and sputum culture conversion are evaluated by time to culture positivity (TTP) in liquid medium system BACTEC MGIT (MGIT, mycobacteria growth indicator tube) 960 of induced sputum samples collected at day 0, 5 and at week 1, 2 and 8 after treatment initiation.

Clinical symptoms are assessed by a clinical scoring tool (TBscore II). Final treatment outcome and occurrence of relapse after the end of treatment are recorded according to World Health Organization (WHO) definitions.

Peak drug concentration (Cmax) and area under the plasma concentration-time curve (AUC) 0-24h will be estimated by non-compartmental analysis and conditions for early therapeutic drug monitoring (TDM) of high-dose RIF/PZA will be explored by model-based analysis.

Primary and main secondary outcomes in the study are the distribution of pharmacokinetics (Cmax, AUC) of high-dose PZA/RIF regimen, safety in terms of incidence of adverse event/severe adverse event (AE/SAE) probably related or related to TB treatment, and drug exposure (AUC) of high-dose PZA/RIF in relation to Mycobacterium tuberculosis (Mtb) drug-susceptibility level (MIC) compared with standard-of-care and suggested literature-derived pharmacokinetic/pharmacodynamic (PK/PD) targets.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years and older
* Confirmed pulmonary TB (positive Mtb culture or positive polymerase chain reaction (PCR) Mtb-complex)
* Intended to start on first-line TB treatment
* HIV negative
* BMI >17
* Written Informed Consent
* Women of childbearing potential should agree on adequate contraceptives during treatment period and have a negative pregnancy test prior to treatment initiation

Exclusion Criteria:

* Not able to provide informed consent/unable to assimilate study information
* Concomitant infectious disease that requires treatment
* Known allergy to rifamycins, isoniazid, pyrazinamide, ethambutol or history of severe sideeffect to any of the drugs
* Drug-induced inflammatory liver diseases in medical history
* History of acute liver disease
* On-going liver disease including hepatitis and elevated transaminase levels >x5 upper normal limit
* Porphyria
* Drug-drug interaction between concomitant drugs and rifampicin that could not be bridged by dose-adjustment of the concomitant drug
* Jaundice
* Acute gout
* Treatment of active TB during the last year
* Drug resistance to RIF, INH, PZA or EMB
* Miliary TB
* Pulmonary TB with smear positivity grade 3 and/or chest X-ray grading equal to advanced TB
* TB in the central nervous system
* Extrapulmonary TB (outside central nervous system) without pulmonary TB
* Pregnancy and breast-feeding
* Immunosuppressive condition
* Heart failure (NYHA class III and IV)
* Renal failure with estimated glomerular filtration rate (eGFR) <50 mL/min
* Dysregulated diabetes mellitus
* Alcohol and drug abuse
* Weight <35 kg or >90 kg
* Participation in other clinical trial (investigating a drug) within the last 30 days prior to study inclusion
* Person who the investigator, after consultation with the central contact persons of the study, finds by other reason than the above listed not suitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) of 40 mg/kg PZA in a high-dose RIF regimen compared with standard-of-care | At treatment Day 14
  PZA AUC(0-24h) at Day 14 after treatment initiation

SECONDARY OUTCOMES:
Safety of 35 mg/kg RIF and 40 mg/kg PZA compared with standard-of-care: AE and SAE | 4 months in the intervention arm, 6 months in the control arm
  Registration of AE/SAE (incidence, severity, drug relatedness, leading to early withdrawal, and leading to death)
Peak Plasma Concentration (Cmax) of 40 mg/kg PZA in a high-dose RIF regimen compared with standard-of-care | At treatment Day 14
  PZA Cmax at Day 14 after treatment initiation
Area under the plasma concentration-time curve (AUC) of high-dose RIF in combination with PZA 40 mg/kg compared with standard-of-care | At treatment Day 14
  RIF AUC(0-24h) at Day 14 after treatment initiation
Peak Plasma Concentration (Cmax) of high-dose RIF in combination with PZA 40 mg/kg compared with standard-of-care | At treatment Day 14
  RIF Cmax at Day 14 after treatment initiation
Drug exposure of PZA 40 mg/kg in relation to Mtb drug-susceptibility level (MIC) compared with standard-of-care and literature-derived suggested PK/PD targets | Day 0 (MIC) and Day 14 (AUC)
  PZA AUC/MIC
Drug exposure of RIF 35 mg/kg in relation to Mtb drug-susceptibility level (MIC) compared with standard-of-care and literature-derived suggested PK/PD targets | Day 0 (MIC) and Day 14 (AUC)
  RIF AUC/MIC
Prediction of PZA pharmacokinetics at steady state (Day 14) based on drug concentration measurement at treatment Day 1 | At treatment Day 1 (first dose) and Day 14
  PZA AUC(0-24h) at Day 1 compared with PZA AUC(0-24h) at Day 14
Prediction of RIF pharmacokinetics at steady state (Day 14) based on drug concentration measurement at treatment Day 1 | At treatment Day 1 (first dose) and Day 14
  RIF AUC(0-24h) at Day 1 compared with RIF AUC(0-24h) at Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Niward, MD, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Linköping University Hospital, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No
Needs additional approval (Amendment) from the Ethical Committee in Sweden.

REFERENCES:
- [Derived] Ekqvist D, Bornefall A, Augustinsson D, Sonnerbrandt M, Nordvall MJ, Fredrikson M, Carlsson B, Sandstedt M, Simonsson USH, Alffenaar JC, Paues J, Niward K. Safety and pharmacokinetics-pharmacodynamics of a shorter tuberculosis treatment with high-dose pyrazinamide and rifampicin: a study protocol of a phase II clinical trial (HighShort-RP). BMJ Open. 2022 Mar 10;12(3):e054788. doi: 10.1136/bmjopen-2021-054788. PMID 35273049